CLINICAL TRIAL: NCT04108832
Title: Traditional Chinese Medicine Formula Liu-Wei-Die-Huang-Wan in the Treatment of Osteoarthritis. An Eight-Weeks Double Blind Randomized Placebo-Controlled Clinical Trial.
Brief Title: Traditional Chinese Medicine Formula Liu-Wei-Die-Huang-Wan in the Treatment of Osteoarthritis.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, Cheng-Chung Wei, Professor, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CS13048
Record Dates: First submitted 2014-09-17; First posted 2019-09-30 (Actual); Last update posted 2019-09-30 (Actual); Status verified 2019-09

CONDITIONS: Osteoarthritis
Keywords: Traditional Chinese Medicine; Herbs; Liu-wei-die-Huang-Wan
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TCM OA2 (Experimental): TCM OA2 3G BID FOR 8 WEEKS
  Interventions: Drug: TCM OA2
- PLACEBO (Placebo Comparator): PLACEBO
  Interventions: Drug: PLACEBO

INTERVENTIONS:
Drug: TCM OA2 — Usage: 3g twice daily
  Other Names: LIOW WEY DIH HUANG WAN EXTRACT PILL
  Arms: TCM OA2
Drug: PLACEBO — Usage: 3g twice daily
  Arms: PLACEBO

SUMMARY:
Through an eight-week randomized, double-blind, placebo-controlled clinical trials formula to evaluate Chinese herbal compound OA2 improve osteoarthritis of efficacy and safety.

DETAILED DESCRIPTION:
This trial was a 8 weeks' randomized, double-blind, placebo-controlled study. The study was approved by the Institutional Review Board of Chung Shan Medical University hospital, and signed informed consent was obtained from each patient. Eighty-one patients of osteoarthritis of knees or hips were enrolled in this study. Inclusion criteria were: age 20 to 80 years; primary osteoarthritis in at least 1 knee, verified radiologically and scored (as normal, minimal, moderate or marked) for joint-space narrowing and marginal osteophytes in the medial, lateral and patellofemoral compartments; at least moderate pain during the 2 weeks before random assignment to treatment, as identified with the Western Ontario and McMaster Universities (WOMAC) LK3.0 Osteoarthritis Index pain subscale.

Primary outcome measures: WOMAC (Western Ontario and McMaster Universities) osteoarthritis index at week 4.

Secondary outcome measures: WOMAC (Western Ontario and McMaster Universities) osteoarthritis index at week 2; Visual analogue scale (VAS), Quality of life by SF-36, patient global assessment (PGA), at week 2 and 4; The PGA was scored from 0 to 4 (0 representing very good); Biomarkers: Hs-CRP, ESR.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥20 years old
* Written informed consent obtained
* Been diagnosed with knee or hip osteoarthritis
* The physician interpretation of X-ray identification and joint space narrowing or bone spurs confirmed
* In randomized trials before entering if used steroids or non-steroid medications osteoarthritis stable doses required at least one week
* The WOMAC osteoarthritis index of the degree of pain assessment in the past two weeks at least> 4ppm pain

Exclusion Criteria:

* Pregnant or breast-feeding women.
* Chemotherapy or radiation therapy in cancer patients

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2012-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities (WOMAC) | week 0, week 4, week 8
  The investigators use WOMAC to compared the difference between the week 8 and week 0

SECONDARY OUTCOMES:
Visual Analog Scale for pain (VAS) | week0, week 4 and 8
  The investigators use VAS to compared the difference between the week 4 and week 0, week 8 and week 0
Physicians Global Assessment to measure quality of life (PGA) | week0, week 4 and week 8
  The investigators use PGA to compared the difference between the week 4 and week 0, week 8 and week 0
Quality of life by SF-36 | week0, week 2 and week 4
  The investigators use SF-36 to compared the difference between the week 4 and week 0, week 2 and week 0
High sensitivity C-reactive protein (Hs-CRP) | week0, week 8
  The investigators use Hs-CRP to compared the difference between the week 8 and week 0
Erythrocyte sedimentation rate (ESR) | week0, week 8
  The investigators use ESR to compared the difference between the week 8 and week 0

CONTACTS AND LOCATIONS:
Overall Officials: Wei C- C, M.D., Study Director — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No